CLINICAL TRIAL: NCT01622868
Title: Phase II Randomized Study of Whole Brain Radiotherapy/Stereotactic Radiosurgery in Combination With Concurrent Lapatinib in Patients With Brain Metastasis From HER2-Positive Breast Cancer - A Collaborative Study of NRG Oncology and KROG
Brief Title: Whole-Brain Radiation Therapy or Stereotactic Radiosurgery With or Without Lapatinib Ditosylate in Treating Patients With Brain Metastasis From HER2-Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01977; NCI-2012-01977 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RTOG-1119; CDR0000735353; RTOG-1119 (Other: NRG Oncology); RTOG-1119 (Other: CTEP); U10CA180868 (NIH); U10CA021661 (NIH)
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: HER2-Positive Breast Carcinoma; Invasive Breast Carcinoma; Metastatic Malignant Neoplasm in the Brain; Recurrent Breast Carcinoma; Stage IV Breast Cancer AJCC v6 and v7
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms | interventions — Lapatinib; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (WBRT or SRS) (Experimental): Patients undergo WBRT 5 days a week for 3 weeks for a total of 15 treatments, or SRS for 1 treatment.
  Interventions: Other: Laboratory Biomarker Analysis; Radiation: Stereotactic Radiosurgery; Radiation: Whole-Brain Radiotherapy
- Arm B (lapatinib ditosylate, WBRT or SRS) (Experimental): Patients undergo WBRT or SRS as in Arm A. Patients also receive lapatinib ditosylate PO QD for 6 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lapatinib Ditosylate; Radiation: Stereotactic Radiosurgery; Radiation: Whole-Brain Radiotherapy

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lapatinib Ditosylate — Given PO
  Other Names: Tykerb
  Arms: Arm B (lapatinib ditosylate, WBRT or SRS)
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
Radiation: Whole-Brain Radiotherapy — Undergo WBRT
  Other Names: WBRT; whole-brain radiation therapy

SUMMARY:
This randomized phase II trial studies how well whole-brain radiation therapy or stereotactic radiosurgery with or without lapatinib ditosylate works in treating patients with breast cancer that has too many of a protein called human epidermal growth factor receptor 2 (HER2) on its cells and has spread to the brain. Radiation therapy uses high energy x rays to kill tumor cells and shrink tumors. Stereotactic radiosurgery is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may kill more tumor cells and cause less damage to normal tissue. Lapatinib ditosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether whole-brain radiation therapy or stereotactic radiosurgery together with lapatinib ditosylate is an effective treatment for brain metastasis from breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if there is a signal for an increase in complete response (CR) rate in the measurable brain metastases at 12 weeks post radiation therapy (RT) (whole brain or stereotactic radiosurgery [SRS]) as determined by magnetic-resonance imaging (MRI) scan of the brain, with the addition of lapatinib (lapatinib ditosylate) to whole-brain radiation therapy (WBRT)/SRS compared to WBRT/SRS alone.

SECONDARY OBJECTIVES:

I. To evaluate CR rate of the measurable brain metastases at 4 weeks post RT (WBRT/SRS) as determined by MRI scan of the brain, with the addition of lapatinib to WBRT/SRS compared to WBRT/SRS alone.

II. To evaluate objective response rate of measurable brain metastases at 4 and 12 weeks post RT (WBRT/SRS) as determined by MRI scan of the brain, with the addition of lapatinib to WBRT/SRS compared to WBRT/SRS alone.

III. To evaluate targeted lesion-specific objective response rate (CR + partial response [PR]) at 4 and 12 weeks post WBRT/SRS.

IV. To evaluate central nervous system (CNS) progressive disease outside the targeted measurable disease with addition of lapatinib to WBRT/SRS compared to WBRT/SRS alone.

V. To evaluate targeted lesion-specific progression at 4 and 12 weeks post WBRT/SRS.

VI. To evaluate treatment related adverse events when adding lapatinib to WBRT/SRS compared to WBRT/SRS alone.

VII. To evaluate overall CNS complete response: disappearance of all CNS target lesions sustained for at least 4 weeks; with no new lesions, no use of corticosteroids, and patient is stable or improved clinically, when adding lapatinib to WBRT/SRS compared to WBRT/SRS alone.

VIII. To evaluate overall CNS progressive disease (within or outside targeted measurable disease) with addition of lapatinib to WBRT/SRS compared to WBRT/SRS alone.

IX. To evaluate overall survival when adding lapatinib to WBRT/SRS compared to WBRT/SRS alone.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients undergo WBRT 5 days a week for 3 weeks for a total of 15 treatments or SRS for 1 treatment.

ARM B: Patients undergo WBRT or SRS as in Arm A. Patients also receive lapatinib ditosylate orally (PO) once daily (QD) for 6 weeks.

After completion of study treatment, patients are followed up at 4 and 12 weeks and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of invasive breast cancer
* HER2-overexpressing breast cancer (3+ staining by immunohistochemistry or HER2 gene amplification by fluorescent in situ hybridization [FISH] or silver in situ hybridization [SISH] >= 2.0)
* At least 1 measurable unirradiated parenchymal brain metastasis within 21 days prior to study entry; patients who are to undergo SRS must have no more than 10 brain metastases; there is no limit on number of brain metastases for WBRT; the minimum size as measured on T1-weighted gadolinium-enhanced MRI must be as follows according to the number of brain metastases:

  * For a single solitary lesion the size must be >= 10 mm
  * For 2 or more lesions, the size of at least 2 of the lesions must be >= 5 mm
  * Patients may also have the following provided the size requirements above are met:

    * Progressive parenchymal brain metastasis following stereotactic radiosurgery for 1-3 brain metastases, with at least 1 new measurable brain lesion
    * Progressive parenchymal brain metastasis following surgical resection of 1-3 brain metastases, with at least 1 measurable brain lesion
* History/physical examination within 21 days prior to study entry
* Karnofsky performance status >= 60 within 21 days prior to study entry
* Able to swallow and retain oral medication (note: for patients unable to swallow tablets, an oral suspension preparation is acceptable)
* Absolute neutrophil count (ANC) >= 1,200 cells/mm^3 (within 21 days prior to study entry)
* Platelets >= 70,000 cells/mm^3 (within 21 days prior to study entry)
* Hemoglobin >= 8.0 g/dL (note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dL is acceptable) (within 21 days prior to study entry)
* Creatinine < 1.5 times institutional upper limit of normal (within 21 days prior to study entry)
* Bilirubin < 1.5 times institutional upper limit of normal (within 21 days prior to study entry)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3.0 times institutional upper limit of normal with or without liver metastasis (within 21 days prior to study entry)
* Patient must provide study specific informed consent prior to study entry
* Women of childbearing potential must have a negative serum pregnancy test within 21 days prior to study entry
* Sexually active women of childbearing potential and sexually active men must practice adequate contraception during therapy and for 12 months after protocol treatment completion
* Prior lapatinib is allowed as long as the last dose received was > 21 days prior to study entry and provided the patient has not received it at any time after the diagnosis of brain metastasis

Exclusion Criteria:

* Prior WBRT
* Prior radiation therapy (RT) (any site) with concurrent lapatinib defined as 1 or more days on which the patient received both radiation therapy and lapatinib on the same day
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Prior invasive malignancy (except non-melanomatous skin cancer, curatively resected thyroid papillary carcinoma, and invasive and non-invasive cancers related to the breast cancer) unless disease free for a minimum of 3 years
* Leptomeningeal disease
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields except patients who have progressed following stereotactic radiosurgery for 1-3 brain metastases, with at least one new lesion
* Severe, active co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of study entry
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of study entry
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; hepatic or biliary disease that is acute or currently active or that requires antiviral therapy (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease per investigator assessment)
  * History of left ventricular ejection fraction (LVEF) below institutional normal unless repeated and within institutional normal range within 90 days of study entry
* Grade 2 or greater rash of any cause at time of study entry
* Grade 2 or greater diarrhea of any cause at time of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: In A Kim, Principal Investigator — NRG Oncology
Locations (302):
- United States (292):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - The Kirklin Clinic at Acton Road, Birmingham, Alabama
  - University of South Alabama Mitchell Cancer Institute, Mobile, Alabama
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Sutter Davis Hospital, Davis, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Mercy General Hospital Radiation Oncology Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Northeast Georgia Medical Center-Gainesville, Gainesville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - UChicago Medicine Comprehensive Cancer Center - Saint Joseph Hospital, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Norton Suburban Hospital and Medical Campus, Louisville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Hospital Niles, Niles, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Renown Regional Medical Center, Reno, Nevada
  - Elliot Hospital, Manchester, New Hampshire
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Mount Sinai Hospital, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Cleveland Clinic Akron General, Akron, Ohio
  - Radiation Oncology Center, Alliance, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Salem Regional Medical Center, Salem, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Jefferson Abington Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
- Canada (2):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Jewish General Hospital, Montreal, Quebec
- South Korea (8):
  - Keimyung University-Dongsan Medical Center, Dalseo-gu, Daegu
  - National Cancer Center-Korea, Goyang-si, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Hwasun-gun, Jeollanam-do
  - Samsung Medical Center, Seoul, Korea
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Gangnam Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System-Severance Hospital, Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Therapy: Stereotactic radiosurgery (SRS) or 3 weeks of whole brain radiotherapy (WBRT)
- Lapatinib and Radiation Therapy: 1000 mg Lapatinib for six weeks with radiation therapy (stereotactic radiosurgery (SRS) or 3 weeks of whole brain radiotherapy (WBRT))
Period: Overall Study
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy
Started | 72 | 71
Eligible | 65 | 71
Eligible, Started Study Treatment, Has Adverse Event Data | 63 | 71
Completed (Participants contributing data to results are considered to have completed the study) | 65 | 71
Not Completed | 7 | 0
Not completed — Protocol Violation | 7 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy | Total
Number analyzed (Participants) | 65 | 71 | 136
Age, Customized [Count of Participants; unit: Participants]
  < 50 years | 22 | 25 | 47
  ≥ 50 years | 43 | 46 | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 71 | 136
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 57 | 67 | 124
  Unknown or Not Reported | 0 | 1 | 1
Karnofsky Performance Status [Count of Participants; unit: Participants] — 60: Requires occasional assistance, but is able to care for most personal needs; 70: Cares for self, unable to carry on normal activity or do active work; 80: Normal activity with effort, some sign or symptoms of disease; 90: Able to carry on normal activity; minor signs or symptoms of disease; 100: Normal, no complaints, no evidence of disease.
  Participants
    60 | 9 | 2 | 11
    70-80 | 29 | 27 | 56
    90-100 | 27 | 42 | 69
Graded Prognostic Assessment for Breast Cancer (Breast-GPA) [Count of Participants; unit: Participants] — Breast-GPA is defined by the combination of prognostic factors: breast tumor subtype, Karnofsky performance score (KPS), and age. Breast tumor subtype consists of the presence/absence of each of the following biomarkers: estrogen receptor, human epidermal growth factor receptor 2, and progesterone receptor. A lower GPA is associated with worse survival; a higher GPA is associated with better survival.
  Participants
    1.5-2.0 | 5 | 4 | 9
    2.5-3.0 | 35 | 37 | 72
    3.5-4.0 | 25 | 30 | 55
Use of Non-central nervous system (CNS) penetrating HER2 Blockade at Study Entry [Count of Participants; unit: Participants] — HER2: human epidermal growth factor receptor 2
  Participants
    No (None) | 23 | 28 | 51
    Yes (Trastuzumab and/or Pertuzumab) | 42 | 43 | 85
Previous Stereotactic SRS or Surgery [Count of Participants; unit: Participants] — Population: Eligible participants randomized before the October 2016 protocol amendment which removed this stratification factor.
  Participants
    number analyzed (Participants) | 42 | 47 | 89
    No | 37 | 41 | 78
    Yes | 5 | 6 | 11
Planned RT [Count of Participants; unit: Participants]
  SRS | 6 | 6 | 12
  WBRT | 59 | 65 | 124

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate in the Brain at 12 Weeks Post-radiation Therapy (RT) Using the RECIST 1.1 Criteria Based on Brain Magnetic Resonance Imaging (MRI)
Description: The Response Evaluation Criteria in Solid Tumors (RECIST) criteria evaluates changes in the largest diameter (unidimensional measurement) of the tumor lesions. Complete response is defined as the complete disappearance of all enhancing disease and off all steroids. Rate is calculated by dividing the number of patients with complete response by the number of analyzable patients.
Time Frame: Baseline and 12 weeks post RT (approximately 12 weeks from start of treatment if SRS and 15 if WBRT)
Population: Evaluable data for determining the 12-week post-RT RECIST response was available for 52 eligible participants on the RT alone arm and 64 on the lapatinib arm.
Measure: Number; unit: percentage of participants
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy
Number analyzed (Participants) | 52 | 64
percentage of participants | 5.8 | 0
Statistical Analysis 1: Comparison: Radiation Therapy vs Lapatinib and Radiation Therapy; The study was designed to see if there is a signal in the 12-week CR rate with the addition of lapatinib to warrant a future phase III trial. Null hypothesis: the 12-week post-WBRT/SRS CR rate is ≤ 5%; alternative hypothesis: the addition of lapatinib will increase that CR rate to at least 20%. 114 eligible participants provide 86% power to detect a 15% absolute increase in CR rate at a significance level of 0.10, using a 1-sided Z-test for the difference of 2 proportions; Test type: Superiority; p = 0.97, Z-test — One-sided significance level = 0.10

2. Secondary Outcome: Complete Response Rate in the Brain at 4 Weeks Post-RT Using the RECIST 1.1 Criteria Based on Brain MRI
Description: The RECIST criteria evaluates changes in the largest diameter (unidimensional measurement) of the tumor lesions. Complete response is defined as the complete disappearance of all enhancing disease and off all steroids. Rate is calculated by dividing the number of patients with complete response by the number of analyzable patients.
Time Frame: Baseline and 4 weeks post RT (approximately 4 weeks from start of treatment if SRS and 7 if WBRT)
Population: Evaluable data for determining the 4-week post-RT RECIST response was available for 55 eligible participants on the RT alone arm and 67 on the lapatinib arm.
Measure: Number; unit: percentage of participants
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy
Number analyzed (Participants) | 55 | 67
percentage of participants | 3.6 | 1.5
Statistical Analysis 1: Comparison: Radiation Therapy vs Lapatinib and Radiation Therapy; Test type: Superiority; p = 0.78, Z-test — One-sided significance level = 0.10

3. Secondary Outcome: Complete Response Rate in the Brain Using the World Health Organization (WHO)/Modified McDonald Criteria Based on Brain MRI
Description: The WHO/modified McDonald Criteria evaluates changes in bidimensional tumor measurements. Complete response is defined as the complete disappearance of all enhancing disease and off all steroids. Rate is calculated by dividing the number of patients with complete response by the number of analyzable patients.
Time Frame: Baseline, 4 and 12 weeks post RT (approximately 4 and 12 weeks from start of treatment if SRS, 7 and 15 if WBRT)
Population: Evaluable data for determining the 4- and 12-week post-RT WHO response was available for 55 eligible participants at week 4 and 52 at week 12 on the RT alone arm and 67 at week 4 and 64 at week 12 on the lapatinib arm.
Measure: Number; unit: percentage of participants
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy
Number analyzed (Participants) | 65 | 71
percentage of participants
  4 weeks post-RT: number analyzed (Participants) | 55 | 67
  4 weeks post-RT | 3.6 | 1.5
  12 weeks post-RT: number analyzed (Participants) | 52 | 64
  12 weeks post-RT | 5.8 | 0
Statistical Analysis 1: Comparison: Radiation Therapy vs Lapatinib and Radiation Therapy; 4 weeks post-RT; Test type: Superiority; p = 0.78, Z-test — One-sided significance level = 0.10
Statistical Analysis 2: Comparison: Radiation Therapy vs Lapatinib and Radiation Therapy; 12 weeks post-RT; Test type: Superiority; p = 0.97, Z-test — One-sided significance level = 0.10

4. Secondary Outcome: Objective Response Rate in the Brain Using the RECIST 1.1 Criteria Based on Brain MRI
Description: The RECIST criteria evaluates changes in the largest diameter (unidimensional measurement) of the tumor lesions. Objective response is defined as a complete or partial response. Complete response is defined as the complete disappearance of all enhancing disease and off all steroids. Partial response is defined as ≥ 30% reduction in the sum of diameters of up to 2 of the largest target lesions. Rate is calculated by dividing the number of patients with objective response by the number of analyzable patients.
Time Frame: Baseline, 4 and 12 weeks post RT (approximately 4 and 12 weeks from start of treatment if SRS, 7 and 15 if WBRT)
Population: Evaluable data for determining the 4- and 12-week post-RT RECIST response was available for 55 eligible participants at week 4 and 52 at week 12 on the RT alone arm and 67 at week 4 and 64 at week 12 on the lapatinib arm.
Measure: Number; unit: percentage of participants
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy
Number analyzed (Participants) | 65 | 71
percentage of participants
  4 weeks post-RT: number analyzed (Participants) | 55 | 67
  4 weeks post-RT | 41.8 | 55.2
  12 weeks post-RT: number analyzed (Participants) | 52 | 64
  12 weeks post-RT | 59.6 | 46.9

5. Secondary Outcome: Percentage of Participants With Progression in the Brain Outside the Targeted Measurable Disease Using the RECIST 1.1 Criteria Based on Brain MRI
Description: The RECIST criteria evaluates changes in the largest diameter (unidimensional measurement) of the tumor lesions. CNS progressive disease outside the targeted measureable disease was determined by a retrospective central review of MRI scans by the study neuroradiology co-chair and is defined as the first occurrence since baseline of new lesions or progression of non-target lesions. Time to CNS progressive disease is defined as time from randomization to the date of progressive disease, last known follow-up (censored), or death (competing risk). Progression rates are estimated using the cumulative incidence method. One-year rates are provided.
Time Frame: From randomization to last follow-up. MRIs occurred at baseline, 4 and 12 weeks post RT, then every 12 weeks thereafter until progression. Maximum follow-up at time of analysis was 71.6 months.
Population: MRI scans were available for central review for progression outside targeted measurable disease for 41 eligible participants on the RT alone arm and 57 on the lapatinib arm.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy
Number analyzed (Participants) | 41 | 57
percentage of participants | 22.0 [10.7 to 35.7] | 37.7 [25.0 to 50.3]

6. Secondary Outcome: Targeted Lesion-specific Objective Response Rate Using the RECIST 1.1 Measurement Criteria Based on Brain MRI
Description: The RECIST criteria evaluates changes in the largest diameter (unidimensional measurement) of the tumor lesions. Objective response is defined as a complete or partial response. Complete response is defined as the complete disappearance of all enhancing disease and partial response is defined as ≥ 30% reduction in the diameter of the target lesion. Lesions were evaluated individually. Rate is calculated by dividing the number of lesions with objective response by the number of analyzable lesions.
Time Frame: Baseline, 4 and 12 weeks post RT (approximately 4 and 12 weeks from start of treatment if SRS, 7 and 15 if WBRT)
Population: Evaluable data for determining the 4- and 12-week post-RT RECIST target lesion measurement response was available for 51 eligible participants at week 4 and 43 at week 12 on the RT alone arm and 66 at week 4 and 57 at week 12 on the lapatinib arm.
Measure: Number; unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy
Number analyzed (Participants) | 65 | 71
Number analyzed (lesions) | 90 | 116
percentage of lesions
  4 weeks post-RT: number analyzed (Participants) | 51 | 66
  4 weeks post-RT | 51.1 | 56.0
  12 weeks post-RT: number analyzed (Participants) | 43 | 57
  12 weeks post-RT: number analyzed (lesions) | 76 | 101
  12 weeks post-RT | 75.0 | 61.4

7. Secondary Outcome: Targeted Lesion-specific Progression Rate Using the RECIST 1.1 Measurement Criteria Based on Brain MRI
Description: The RECIST criteria evaluates changes in the largest diameter (unidimensional measurement) of the tumor lesions. Progression is defined as ≥ 20% increase in the diameter of the target lesion relative to nadir. Lesions were evaluated individually. Rate is calculated by dividing the number of lesions with progression by the number of analyzable lesions.
Time Frame: Baseline, 4 and 12 weeks post RT (approximately 4 and 12 weeks from start of treatment if SRS, 7 and 15 if WBRT)
Population: as for outcome 6
Measure: Number; unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy
Number analyzed (Participants) | 65 | 71
Number analyzed (lesions) | 90 | 116
percentage of lesions
  4 weeks post-RT: number analyzed (Participants) | 51 | 66
  4 weeks post-RT | 3.3 | 1.7
  12 weeks post-RT: number analyzed (Participants) | 43 | 57
  12 weeks post-RT: number analyzed (lesions) | 76 | 101
  12 weeks post-RT | 6.6 | 14.9

8. Secondary Outcome: Frequency of Highest Treatment-related Adverse Event Per Participant
Description: Adverse events reported as definitely, probably, or possibly related to protocol treatment. Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death. Summary data provided in this outcome measure. See Adverse Events Module for specific Adverse Event data.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 71.6 months.
Population: Eligible participants who started study treatment and have adverse event data.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy
Number analyzed (Participants) | 63 | 71
Participants
  Grade 1 | 8 | 14
  Grade 2 | 23 | 20
  Grade 3 | 5 | 20
  Grade 4 | 0 | 4
  Grade 5 | 0 | 0

9. Secondary Outcome: Overall Complete Response Rate in the Brain Using the RECIST 1.1 Criteria Based on Brain MRI
Description: The RECIST criteria evaluates changes in the largest diameter (unidimensional measurement) of the tumor lesions. Overall complete response is defined as the complete disappearance of all CNS target lesions sustained for at least 4 weeks; with no new lesions, no use of corticosteroids, and patient is stable or improved clinically. All site-reported MRI data and all site-reporting of clinical progressive disease indicators were used in this analysis. Rate is calculated by dividing the number of participants with overall complete response by the number of analyzable participants.
Time Frame: as for outcome 5
Population: Evaluable data for determining overall post-RT RECIST response was available for 54 eligible participants on the RT alone arm and 68 on the lapatinib arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy
Number analyzed (Participants) | 54 | 68
Participants | 0 | 0
Statistical Analysis 1: Comparison: Radiation Therapy vs Lapatinib and Radiation Therapy; Test type: Superiority; p = 1.00, z-test — One-sided significance level = 0.10

10. Secondary Outcome: Overall Progression Rate in the Brain Using the RECIST 1.1 Criteria Based on Brain MRI
Description: The RECIST criteria evaluates changes in the largest diameter (unidimensional measurement) of the tumor lesions. Overall progression is defined as unequivocal progression, new or worsening tumor-related neurological symptoms, tumor-related increase in steroid dose, new primary in brain, or progression in target lesions. All site-reported MRI data and all site-reporting of clinical progressive disease indicators were used in this analysis. Rate is calculated by dividing the number of participants with progression by the number of analyzable participants.
Time Frame: as for outcome 5
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy
Number analyzed (Participants) | 54 | 68
Participants | 38 | 54

11. Secondary Outcome: Overall Survival (OS)
Description: An event for overall survival is death due to any cause. Survival time is defined as time from randomization to the date of death or last known follow-up (censored). Rates are estimated by the Kaplan-Meier method. Analysis occurred after 101 deaths were reported.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 71.6 months.
Population: Eligible participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy
Number analyzed (Participants) | 65 | 71
months | 15.6 [8.4 to 19.1] | 15.3 [12.3 to 21.0]
Statistical Analysis 1: Comparison: Radiation Therapy vs Lapatinib and Radiation Therapy; Test type: Superiority; p = 0.67, Log Rank — Two-sided significance level = 0.05; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.62 to 1.36]

ADVERSE EVENTS:
Time Frame: Weekly during radiation therapy and lapatinib (when applicable), 4 weeks post-RT completion, 12 weeks post-RT completion, every 3 months to year 3, and then annually. Maximum follow-up at time of analysis was 71.6 months.
Arm/Group | Radiation Therapy | Lapatinib and Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 48/63 | 53/71
Serious Adverse Events (participants affected / at risk) | 17/63 | 16/71
Other Adverse Events (participants affected / at risk) | 49/63 | 63/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy (N=63) | Lapatinib and Radiation Therapy (N=71)
Anemia (Blood and lymphatic system disorders) | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 1 | 1
Fever (General disorders) | 1 | 1
Gait disturbance (General disorders) | 2 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0
Endocarditis infective (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 2
Alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 3
White blood cell decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Nail loss (Skin and subcutaneous tissue disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 2
Vascular disorders - Other, specify (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy (N=63) | Lapatinib and Radiation Therapy (N=71)
Anemia (Blood and lymphatic system disorders) | 5 | 18
Blurred vision (Eye disorders) | 7 | 9
Eye disorders - Other, specify (Eye disorders) | 2 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 5 | 11
Diarrhea (Gastrointestinal disorders) | 5 | 31
Dry mouth (Gastrointestinal disorders) | 3 | 6
Dyspepsia (Gastrointestinal disorders) | 3 | 8
Mucositis oral (Gastrointestinal disorders) | 1 | 9
Nausea (Gastrointestinal disorders) | 16 | 38
Vomiting (Gastrointestinal disorders) | 11 | 21
Edema limbs (General disorders) | 4 | 9
Fatigue (General disorders) | 27 | 40
Gait disturbance (General disorders) | 4 | 11
Pain (General disorders) | 10 | 7
Urinary tract infection (Infections and infestations) | 1 | 4
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 5
Fall (Injury, poisoning and procedural complications) | 1 | 7
Alanine aminotransferase increased (Investigations) | 2 | 12
Alkaline phosphatase increased (Investigations) | 1 | 8
Aspartate aminotransferase increased (Investigations) | 1 | 10
Blood bilirubin increased (Investigations) | 1 | 9
Lymphocyte count decreased (Investigations) | 3 | 17
Platelet count decreased (Investigations) | 3 | 12
Weight loss (Investigations) | 3 | 7
White blood cell decreased (Investigations) | 1 | 11
Anorexia (Metabolism and nutrition disorders) | 12 | 19
Dehydration (Metabolism and nutrition disorders) | 0 | 5
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 11
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 7
Hypokalemia (Metabolism and nutrition disorders) | 0 | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 4
Hyponatremia (Metabolism and nutrition disorders) | 2 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 8
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 12
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 6 | 6
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4
Ataxia (Nervous system disorders) | 3 | 4
Cognitive disturbance (Nervous system disorders) | 4 | 2
Dizziness (Nervous system disorders) | 7 | 19
Dysarthria (Nervous system disorders) | 1 | 4
Dysgeusia (Nervous system disorders) | 3 | 9
Headache (Nervous system disorders) | 21 | 27
Lethargy (Nervous system disorders) | 0 | 4
Memory impairment (Nervous system disorders) | 11 | 9
Nervous system disorders - Other, specify (Nervous system disorders) | 4 | 2
Paresthesia (Nervous system disorders) | 5 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 10
Seizure (Nervous system disorders) | 2 | 5
Anxiety (Psychiatric disorders) | 2 | 8
Confusion (Psychiatric disorders) | 2 | 6
Depression (Psychiatric disorders) | 3 | 10
Insomnia (Psychiatric disorders) | 3 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 13
Alopecia (Skin and subcutaneous tissue disorders) | 19 | 24
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 7
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 | 5
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 5
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 18
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 10
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 | 7
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 4
Hypertension (Vascular disorders) | 2 | 11
Lymphedema (Vascular disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior approval from the sponsor. In addition, PI's are required to abide by the collaborator's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT01622868/Prot_SAP_000.pdf